CLINICAL TRIAL: NCT01937286
Title: Single Center Experience Over a Decade in Living Donor Liver Transplantation for Egyptian Patients With Hepatocellular Carcinoma: Stretching the Limits
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of Tropical Medicine, Ain Shams University
Other Study IDs: Hepatocellular carcinaoma
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Recurrence of HCC After LDLT
Keywords: LDLT,HCC, Microvascular invasion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Within community with high incidence of HCC, stretching the limits could be justified based on tumor characters and its biological behavior

DETAILED DESCRIPTION:
590 Egyptian patients underwent LDLT; of them, 172 (32%) patients were transplanted for HCC. Twenty six cases (15.1%) were excluded due to early postoperative mortality (n=22) or due to non HCC related mortality (n=4). One hundred forty six patients were retrospectively reviewed to determine prognostic factors for recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Egyptien Patients with HCC
* Patients within Milan Criteria
* Patients beyond Milan criteria are selected on a case by case basis until 2005. From 2005 , patients beyond Milan criteria are subjected to down staging protocol and then reassessed (pre transplantation local ablative therapy either with RFA or TACE according to the size and the site of the lesion and we wait for 12 weeks after ablation ,only those with well ablated lesions, decreased AFP and no denovo lesions were transplanted).

Exclusion Criteria:

* • Evidence of macro vascular invasion by CT portography and/or US duplex.

  * Metastatic HCC
  * General contraindications for LT (ongoing sepsis, other major co morbidities,…).
  * Early postoperative mortality (first1 month).
  * Post transplant mortality during the period of follow up due to any cause other than recurrent HCC (e.g. sepsis, rejection, cardiological or cerebrovascular complications…)

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyptien Patient with HCC who underwent LDLT
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2002-01; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Recurrence of Hepatocellular carcinoma after LDLT | at least 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Center For Organ Transplantation (ASCOT),Ain Shams university, Cairo, Egypt